CLINICAL TRIAL: NCT06355310
Title: Mechanisms of SGLT2 Inhibition in Pediatric Steatotic Liver Disease
Acronym: SHIELD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Justin Ryder (Other)
Responsible Party: Sponsor-Investigator, Justin Ryder, Vice Chair of Research for the Department of Surgery at Ann & Robert H Lurie Children's Hospital, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 2023-6429
Record Dates: First submitted 2024-04-01; First posted 2024-04-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin; Control Groups

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind placebo control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study intervention (Experimental): Empagliflozin 10 mg will be taken daily
  Interventions: Drug: Empagliflozin 10 MG
- Control arm (Placebo Comparator): Placebo oral tablet will be taken daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Participants will take a 10 mg oral tablet of empagliflozin, an orally-active inhibitor of sodium-glucose co-transporter 2 (SGLT2)
  Other Names: Jardiance
  Arms: Study intervention
Drug: Placebo Oral Tablet — Participants will take an identical appearing oral tablet with zero active ingredient.
  Other Names: Control group
  Arms: Control arm

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial specifically designed to evaluate the preliminary feasibility, initial efficacy and safety of SGLT2 inhibitors for treating NAFLD in adolescents with obesity.

DETAILED DESCRIPTION:
The overall aim of this pilot study is to evaluate the feasibility and obtain a preliminary estimate of efficacy and safety of the SGLT2 inhibitor, empagliflozin, in adolescents with obesity (BMI-percentile ≥95th) who have MRI-confirmed NAFLD (hepatic fat fraction ≥ 5.5%) and have normal fasting glucose.

Participants will take empagliflozin, once daily, in the morning, with or without food, in addition to receiving lifestyle/behavioral counseling throughout the study.

The following data will be collected throughout the course of the study: Physical exam with tanner staging, safety and fasting labs, fasting blood draw (biomarkers), urine sample, 2-stage clamp (overnight Stay),Stable isotope tracers (overnight Stay), MRI scan (MRS-Liver), BMI/anthropometrics, urine pregnancy test for female participants, iDXA scan (body fat and bone density), arterial stiffness and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

For clinical referral to screening visit:

* BMI >30 kg/m2 or >95th BMI-Percentile
* Weight Range of 75kg to 150kg
* Age 16 to <21 at baseline
* Elevated alanine aminotransferase (ALT) more than twice the upper limit of normal by gender (≥ 44 U/L for girls, ≥ 50 U/L for boys)63 within 3 months prior to screening (used for historic ALT value) OR diagnosis of NAFLD from ultrasound, MRI, or participants with biopsy-proven NASH within 12 months of screening.
* History of lifestyle modification to treat obesity or NAFLD.
* Tanner stage >2
* Normal fasting glucose (fasting blood glucose <100 mg/dL)

To be obtained at screening visit:

* Confirmation of obesity;
* Tanner stage 2,3,4 or 5;
* Normal fasting glucose tolerance (fasting blood glucose <100 mg/dL);
* If Screening ALT is used as inclusion criteria (if > 2x historic ALT value (historical value obtained clinically within 12 months of screening visit), repeated after 4 weeks [unable to randomize until completed]. If the repeat ALT is more than 50% increased or decreased over the screening ALT, a third ALT should be obtained. If a third ALT is not within 50% of the previous value, then the subject is ineligible but may be rescreened at a later date. If ALT is not used:

  * An ultrasound will be done to diagnose NAFLD if the diagnosis has not previously been made by ultrasound, MRI or biopsy.
  * A MRI-derived HFF ≥ 5.5%
* Willingness to adhere to lifestyle considerations throughout the study

Exclusion Criteria:

* ALT > 250U/L at screening
* History of significant alcohol intake or current use
* Impaired fasting glucose (>100 mg/dL)
* Diabetes (type 1 or 2)
* Current or recent (<6 months prior to enrollment) use of weight loss medication(s)
* Vitamin E supplementation or use of metformin

  -washout period 30 days
* Previous bariatric surgery
* Prior use of empagliflozin
* Lower limb infection/ulceration within 3 months of screening
* Metal or magnetic implants, devices or objects inside of or on the body, which are not MRI compatible
* Structural and functional urogenital abnormalities, that predispose for urogenital infections
* Recent initiation (<3 months prior to enrollment) of anti-hypertensive or lipid medication(s)
* Major psychiatric disorder
* Known hypothalamic or pituitary dysfunction
* Current pregnancy or plans to become pregnant
* Females unwilling to be tested for pregnancy
* Females who are sexually active and not protects by an effective method of birth control (e.g. UID or medication or patch)

  -can re-screen 30 days after getting on birth control
* Tobacco use
* Significant liver dysfunction (levels >5 times the upper limit of normal (ULN)):
* ALT (ULN = 50 U/L)
* AST (ULN = 48 U/L)
* GGT (ULN = 48 U/L)
* ALP (ULN = 115 U/L)
* Platelets < 150,000 cells/mm3
* Total bilirubin > 1.3 mg/dL
* INR > 1.3
* Albumin <3.2 g/dL
* Gilbert's Syndrome
* Any known causes of liver disease (except NAFLD and NASH)
* Significant renal dysfunction (estimated glomerular filtration rate [eGFR] < 80 mL/min/1.73 m2),
* Diagnosed monogenic obesity
* History of cancer
* Untreated thyroid disorder
* History of decompensation events (ascites, variceal bleeding, hepatic encephalopathy, or hepatocellular carcinoma)
* Current or recent (<6 months prior to enrollment) use of medication(s) associated with weight gain (e.g. atypical anti-psychotics).

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Hepatic Fat | 26-Weeks
  change in hepatic fat fraction (Hepatic fat will be measured by MRI via proton density fat fraction (PDFF)) from baseline (first measurement time point) to 26-weeks.

SECONDARY OUTCOMES:
Body mass index | 26-Weeks
  * BMI
  * body fat% (total and visceral fat)
  * ALT
  * biomarkers of NAFLD oCK-18 ototal and activated PAI-1 oIL-8
  * biomarkers of bone health (additional safety outcome) oN-terminal collagen type I extension propeptide (PINP) oOsteocalcin oC-terminal cross-linking telopeptide of type I collagen (CTX)
  * Systolic and diastolic blood pressure
  * glycemic control (from oral glucose tolerance test)
  * Insulin sensitivity (from oral glucose tolerance test) by the whole-body insulin sensitivity index

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ryder, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States